CLINICAL TRIAL: NCT06425003
Title: Mass Balance Study of [14C] ABBV-CLS-7262 in Healthy Male Volunteers Following Single Oral Dose Administration
Brief Title: Study of [14C] ABBV-CLS-7262 in Healthy Male Volunteers Following Single Oral Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calico Life Sciences LLC (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M24-326
Record Dates: First submitted 2024-05-06; First posted 2024-05-22 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C] ABBV-CLS-7262 (Experimental): Participants will receive [14C] ABBV-CLS-7262 on Day 1.
  Interventions: Drug: [14C] ABBV-CLS-7262

INTERVENTIONS:
Drug: [14C] ABBV-CLS-7262 — Oral Solution

SUMMARY:
The purpose of this study is to evaluate mass balance, pharmacokinetics and safety of [14C] ABBV-CLS-7262 in healthy, male volunteers following administration of a single oral dose.

ELIGIBILITY:
Inclusion Criteria:

* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.
* Body Max Index (BMI) is ≥ 18.0 to ≤ 32.0 kg/m2 after rounding to the tenths decimal at screening.

Exclusion Criteria:

* Considering fathering a child or donating sperm during the study and for 94 days after study drug administration, or is unwilling to comply with protocol recommended contraception recommendations.
* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), endocrine, metabolic, renal, hepatic, gastrointestinal, hematologic, endocrinologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* Has had significant exposure to radiation for professional or medical reasons (e.g., serial x-rays or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring), except dental x-rays, within 12 months prior to study drug administration.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 30 days from last dose.
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Maximum observed concentration (Cmax) | Up to approximately Day 15 from last dose
  Cmax will be assessed.
Time to Cmax (peak time, Tmax) | Up to approximately 15 days from last dose
  Tmax will be assessed.
Terminal phase elimination half-life (t1/2) | Up to approximately 15 days from last dose
  Terminal phase elimination half-life (t1/2) will be assessed.
Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable concentration (AUCt) | Up to approximately 15 days from last dose
  AUCt will be assessed.
Percent radioactivity excreted | Up to approximately 15 days from last dose
  Percentage total radioactivity
Identification of metabolites excreted | Up to approximately 15 days from last dose
  Identification of the major metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- Fortrea Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No